CLINICAL TRIAL: NCT00335439
Title: Effect of Prophylactic NSAID Drops on Cystoid Macular Edema After Cataract Surgery Using Optical Coherence Tomography
Brief Title: Effect of Prophylactic Ketorolac on CME After Cataract Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University (Other)
Responsible Party: Principal Investigator, Dr. Sherif R El-Defrawy, Principal Investigator, Queen's University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: QUEENS-SRE-2
Record Dates: First submitted 2006-06-08; First posted 2006-06-09 (Estimated); Last update posted 2016-01-13 (Estimated); Status verified 2016-01

CONDITIONS: Macular Edema, Cystoid
MeSH Terms: conditions — Macular Edema | interventions — Ketorolac Tromethamine

INTERVENTIONS:
Drug: ketorolac tromethamine 0.5% (Acular®)

SUMMARY:
The study will evaluate the efficacy of prophylactic administration of the topical nonsteroidal anti-inflammatory drug (NSAID) ketorolac tromethamine 0.5% (Acular®) on cystoid macular edema (CME) in patients having undergone cataract surgery. CME is the most frequent cause of decreased vision after uncomplicated cataract surgery and can result in irreversible sight reduction. The investigation will involve a comparison arm and a treatment arm with both sets of patient populations being evaluated for CME with ophthalmologic examinations and optical coherence tomography (OCT) measurements. The objective is to elucidate the role of NSAID drops in preventing CME after cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

* First cataract surgery (i.e., first eye).

Exclusion Criteria:

* hypersensitivity to the NSAID drug class,
* pregnancy.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2006-06; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Degree of cystoid macular edema by means of OCT (total macular volume) measurements

CONTACTS AND LOCATIONS:
Overall Officials: Sherif El-Defrawy, MD PhD FRCSC, Principal Investigator — Hotel Dieu Hospital, Kingston General Hospital, Queen's University
Locations (1):
- Hotel Dieu Hospital, Kingston, Ontario, Canada